CLINICAL TRIAL: NCT02327286
Title: Prevenção do Diabetes em Mulheres Com Diabetes Gestacional prévio: Estudo multicêntrico de mudanças Intensivas de Estilo de Vida: LINDA-Brasil
Brief Title: Randomized Clinical Trial of Lifestyle Interventions to Prevent Diabetes in Women With Previous Gestational Diabetes
Acronym: LINDA-Brasil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Eli Lilly and Company (Industry); Hospital de Clinicas de Porto Alegre (Other); Fundação Médica do Rio Grande do Sul (Unknown); Federal University of Pelotas (Other); Centro de Estudos em Diabetes e Hipertensão (Unknown)
Responsible Party: Principal Investigator, MSchmidt, Associate Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 563942/2010-0; U1111-1165-0608 (Registry Identifier: REBEC); 00914312.0.1001.5327 (Registry Identifier: Plataforma Brasil)
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus; Diabetes, Gestational
Keywords: Diabetes Mellitus; Gestational diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes, Gestational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Promote and support healthy behaviors
  Interventions: Behavioral: Promote and support healthy behaviors
- Control (No Intervention): Conventional care for women with prior GDM.

INTERVENTIONS:
Behavioral: Promote and support healthy behaviors — * Exclusive breastfeeding for 6 months and partial breastfeeding for at least 3 additional months.
  * Personally monitored weight loss and maintenance with goal: return to pre-pregnancy weight and, if overweight pre-pregnancy, loss of an additional 5% of body weight.
  * Healthy eating: avoidance of ultra-processed foods, limited intake of oils, sugars and processed foods, increased intake of foodstuffs in their natural state, regular intake of water, dairy products, unsweetened coffee and tea.
  * A progressive increase in physical activity of at least 150 minutes of moderate or vigorous physical activity/week (7500 steps/day) and reduction of sedentary behavior with monitoring by personally worn devices.
  Arms: Intervention

SUMMARY:
Randomized trial aiming to investigate the effectiveness of a lifestyle intervention program implemented within the first year after a pregnancy complicated by gestational diabetes (GDM), in delaying or preventing the development of type 2 diabetes.

DETAILED DESCRIPTION:
LINDA-Brasil is a multicenter randomized clinical trial to test the effectiveness of a lifestyle intervention program tailored to women with a recent diagnosis of GDM to be implemented within two-year after pregnancy with the goal of preventing type 2 diabetes. It is based on a cohort study of women recruited during pregnancy. At first contact, the study protocol is explained, and it is made clear that not all women enrolled in the cohort will be eligible to participate in the post partum clinical trial. During pregnancy and the immediate post-partum period, women are monitored monthly by telephone to maintain contact. From six weeks to two years after delivery, high risk status is determined and women at high risk are contacted to evaluate their eligibility for the trial. Those potentially eligible are then invited to the research center for an examination prior to randomization. Once eligibility is confirmed, women return to the clinical research center at which point key aspects of the clinical trial protocol are reviewed and remaining questions clarified. Those willing to participate provide specific informed consent and are then allocated to one of the two comparison groups. The randomization scheme is 1:1 by trial arm, stratified by center and has random blocks. Based on results of key previous clinical trials on diabetes prevention, LINDA has tailored its intervention to meet the particular needs of women with previous GDM during their post partum. Building from social cognitive theory, interventions are participant-centered, allowing adaptation to each women´s setting, within the limits of a standardized prevention program with defined goals and structure. Communication strategies are based on motivational interviewing and health coaching approaches that can be implemented in the primary care setting. Follow-up is planned to continue until all women have completed at least 18 months of participation and the average length of follow up for the whole sample is at least three years. Outcomes are assessed at baseline, at 6 months and then annually. Women who develop diabetes will be notified and oriented to seek medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or older having gestational diabetes, regardless of the diagnostic criteria, who used insulin during their pregnancy or were found to have impaired glucose tolerance or impaired fasting glucose (>=100 mg/dL) on a post-partum oral glucose tolerance test (OGTT).
* We amended the protocol to also include women using oral hypoglycemics during pregnancy because their use increased during the trial implementation.

Exclusion Criteria:

* Confirmed postpartum diabetes (two abnormal OGTTs) or current use of antidiabetic medication
* Indication that the trial interventions will not be feasible, for example, distance from the trial site
* Poor attendance/response in previous contacts (appointments or phone interviews)
* Health limitations or treatments (assessed by questionnaire) restricting the nutritional intervention or the ability to practice physical activity, affecting glucose tolerance or limiting participation or survival.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Incident diabetes mellitus | Up to 5 years
  Diabetes mellitus as ascertained by a 75g oral glucose tolerance test.

SECONDARY OUTCOMES:
Weight at one year post randomization | 1 year
  Return to pre-pregnancy weight; if overweight or obese before pregnancy, achieve an additional reduction of at least 5%;
  Difference in weight determined between measured weight at 1 year post randomization and self-reported pre-pregnancy weight.

CONTACTS AND LOCATIONS:
Overall Officials: Maria I Schmidt, MD, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (3):
- Brazil (3):
  - Centro de Estudos em Diabetes e Hipertensão, Fortaleza, Ceará
  - Federal University of Pelotas, Pelotas, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul

REFERENCES:
- [Background] Schmidt MI, Duncan BB, Castilhos C, Wendland EM, Hallal PC, Schaan BD, Drehmer M, Costa E Forti A, Facanha C, Nunes MA. Lifestyle INtervention for Diabetes prevention After pregnancy (LINDA-Brasil): study protocol for a multicenter randomized controlled trial. BMC Pregnancy Childbirth. 2016 Mar 30;16:68. doi: 10.1186/s12884-016-0851-x. PMID 27029489
- [Derived] Schmidt MI, Bracco PA, Nunes MA, Cherubini KA, Castilhos CD, Spagiari JZ, Galliano LM, Ladwig R, Del Vecchio FB, Del Vecchio AHM, Drehmer M, Forti AC, Facanha C, Zajdenverg L, de Almeida-Pititto B, Rea RR, Dualib PM, Duncan BB. Telephone lifestyle intervention to prevent diabetes in women with recent gestational diabetes mellitus attending the national health system: the LINDA-Brasil clinical trial. BMJ Open. 2024 Oct 15;14(10):e082572. doi: 10.1136/bmjopen-2023-082572. PMID 39414286
- [Derived] Dame P, Cherubini K, Goveia P, Pena G, Galliano L, Facanha C, Nunes MA. Depressive Symptoms in Women with Gestational Diabetes Mellitus: The LINDA-Brazil Study. J Diabetes Res. 2017;2017:7341893. doi: 10.1155/2017/7341893. Epub 2017 Jun 8. PMID 28685151
- See also: Study protocol — http://bmcpregnancychildbirth.biomedcentral.com.libproxy.lib.unc.edu/articles/10.1186/s12884-016-0851-x